CLINICAL TRIAL: NCT07348497
Title: The Effect of Preoperative Education on Preoperative Anxiety and Emergence Agitation: A Randomized Controlled Trial
Brief Title: Effects of Preoperative Education on Anxiety and Emergence Agitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, İnci Kırtıl, Assistant Professor, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 553868
Record Dates: First submitted 2025-12-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Preoperative Anxiety; Emergence Agitation; Surgical Patients
Keywords: emergence agitation; anxiety; pain
MeSH Terms: conditions — Emergence Delirium; Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Preoperative Emergence-Focused Education (Experimental): Participants in this group will receive routine perioperative care plus a structured, nurse-led preoperative education program focused on the anesthesia emergence process. The education includes information on general anesthesia, endotracheal intubation and extubation, the post-anesthesia care unit environment, and expected physical, emotional, and behavioral responses during emergence. Education is delivered individually in a face-to-face session lasting approximately 10-15 minutes and is supported by written educational materials.
  Interventions: Behavioral: Preoperative Emergence-Focused Education
- Control Group: Standard Perioperative Care (Active Comparator): Participants in this group will receive routine preoperative and perioperative care in accordance with institutional clinical practice, including standard verbal information about the surgical and anesthesia process, without additional emergence-focused education.
  Interventions: Other: Standard Perioperative Care

INTERVENTIONS:
Behavioral: Preoperative Emergence-Focused Education — A standardized preoperative educational intervention delivered by trained nurses to increase patients' understanding of the anesthesia emergence process and to reduce preoperative anxiety and postoperative emergence agitation. The intervention is provided before surgery through verbal education and written materials.
  Arms: Experimental Group: Preoperative Emergence-Focused Education
Other: Standard Perioperative Care — Routine perioperative care provided according to institutional standards, including standard preoperative verbal information.
  Arms: Control Group: Standard Perioperative Care

SUMMARY:
This randomized controlled trial aims to evaluate the effect of structured preoperative education focused on the anesthesia emergence process on preoperative anxiety and postoperative emergence agitation in adult surgical patients undergoing general anesthesia. Emergence agitation is a frequent postoperative complication associated with patient discomfort, safety risks, and increased clinical workload. Preoperative anxiety is considered a modifiable risk factor for emergence agitation; however, evidence-based educational interventions targeting the emergence phase are limited.

The intervention consists of a standardized, nurse-led preoperative education program providing information on general anesthesia, endotracheal intubation and extubation, the post-anesthesia care unit environment, and expected physical and emotional responses during emergence. Education is delivered through a face-to-face individual session supported by written materials. Patients in the control group receive routine perioperative verbal information in accordance with standard care.

Eligible adult patients scheduled for elective general surgery under general anesthesia will be randomly assigned to either the intervention or control group. Preoperative anxiety will be assessed using the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Emergence agitation will be evaluated in the post-anesthesia care unit using the Riker Sedation-Agitation Scale (SAS) and the Richmond Agitation-Sedation Scale (RASS) during the first 30 minutes after surgery.

The primary outcomes are preoperative anxiety levels and the incidence of postoperative emergence agitation. Secondary outcomes include postoperative pain, extubation time and quality, and length of stay in the post-anesthesia care unit. This study seeks to determine whether emergence-focused preoperative education can improve perioperative psychological outcomes and enhance patient safety in surgical care.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to systematically evaluate the effect of structured preoperative education focused on the anesthesia emergence process on preoperative anxiety and postoperative emergence agitation in adult surgical patients undergoing general anesthesia. Emergence agitation is a common and clinically significant phenomenon in the immediate postoperative period and is associated with patient distress, safety risks, increased workload for healthcare professionals, and potential complications. Preoperative anxiety has been identified as a key modifiable risk factor contributing to emergence agitation; however, evidence-based educational interventions specifically targeting the emergence phase remain limited. The intervention consists of a standardized, nurse-led preoperative education program that provides patients with detailed information about the anesthesia emergence process. Educational content includes explanations of general anesthesia, endotracheal intubation and extubation procedures, the physical environment of the post-anesthesia care unit (PACU), expected physiological, emotional, and behavioral responses during emergence, and the typical duration and monitoring of the recovery process. Education is delivered in a face-to-face individual session lasting approximately 10-15 minutes and is supported by a written patient education brochure to ensure consistency and comprehension. Participants will be adult patients (≥18 years) scheduled for elective general surgery under general anesthesia at a tertiary training and research hospital. Eligible patients who provide informed consent and meet inclusion criteria will be randomly assigned to either the intervention group or the control group. Randomization will be performed using a computer-generated random sequence. The control group will receive routine perioperative verbal information in accordance with standard clinical practice, while the intervention group will receive routine care plus the structured emergence-focused education. Preoperative anxiety will be assessed on the day of surgery prior to anesthesia induction using the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Postoperative emergence agitation will be evaluated in the PACU using the Riker Sedation-Agitation Scale (SAS) and the Richmond Agitation-Sedation Scale (RASS). Agitation assessments will be conducted at 10-minute intervals during the first 30 minutes following admission to the PACU, and the highest recorded score will be used for analysis. Emergence agitation will be defined as a SAS score ≥5 and/or a RASS score ≥+1. The primary outcomes of the study are the incidence and severity of emergence agitation and preoperative anxiety levels. Secondary outcomes include maximum postoperative pain scores in the PACU, time to extubation, extubation quality, and length of stay in the PACU. Demographic, clinical, and perioperative variables will be collected using a structured patient information form.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled for elective general surgery under general anesthesia
* American Society of Anesthesiologists (ASA) physical status I-III
* Able to comprehend the educational intervention
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of neurological disorders, cognitive impairment, or dementia
* Severe psychiatric illness or current use of antipsychotic medications
* Alcohol or substance use disorder
* Sensory impairments (visual, hearing, or speech) that may interfere with communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Emergence Agitation | First 30 minutes after admission to the post-anesthesia care unit (PACU)
  Patients' emergence agitation will be assessed using the Riker Sedation-Agitation Scale (SAS) and the Richmond Agitation-Sedation Scale (RASS). Patients with a maximum SAS score ≥5 and RASS score ≥ +1 will be considered positive agitation (the highest score within the first 30 minutes will be taken into account).
Preoperative Anxiety Level | On the day of surgery, prior to induction of anesthesia
  Patients' preoperative anxiety will be assessed using the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Higher scores on the scale will be considered indicative of increased anxiety.

SECONDARY OUTCOMES:
Postoperative Pain Intensity | First 30 minutes after admission to the PACU
  Patients' pain intensity will be assessed using an 11-point numerical rating scale. A score of 0 will indicate that the patient has no pain at all, while a score of 10 will indicate the most severe pain experienced to date. The highest pain score recorded within the first 30 minutes will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan 2.Abdul Hamid Khan Educational and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and confidentiality.